CLINICAL TRIAL: NCT01304667
Title: Chemo- and Radiotherapy in Epithelial Vulvar Cancer
Acronym: CARE
Status: Completed | Type: Observational
Sponsor: AGO Study Group (Other)
Collaborators: medac GmbH (Industry); Philipps University Marburg (Other)
Responsible Party: Sponsor
Other Study IDs: AGO-VOP.1 / CARE
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2015-12

CONDITIONS: Radio/Chemotherapy in Node Positive Advanced Vulvar Cancer
Keywords: Vulvar cancer; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Subproject of Translational Research:
  Paraffin embedded tissue samples were collected.
Oversight: Data Monitoring Committee: No

SUMMARY:
This retrospective, multicenter study is designed to collect tumor characteristics as well as treatment data from patients diagnosed with primary or recurrent squamous cell cancer of the vulva with emphasis on indication and application of radio- and chemotherapy. Application of chemotherapy in primary treatment of vulvar cancer is rare; the study collective is therefore extended to relapsed disease.

DETAILED DESCRIPTION:
All patients with primary squamous cell cancer of the vulva > stage Ia who were diagnosed and received treatment between 1998 and 2008 at the participating centres will be included in the study. Furthermore patients with recurrent disease diagnosed and treated at the participating centres during the same time period can be included given that they not only underwent surgical excision for treatment.

For centers with restricted resources for data entry an alternative study collective was defined:

All Patients with primary or relapsed squamous cell vulvar cancer receiving radio- and/or chemotherapy for treatment at the participating centres between 1998 and 2008 will be included in the study. This also includes node negative patients receiving radio/chemotherapy for other reasons.

The participating centers themselves have to decide which study collective they are documenting, dependent on their available resources.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary squamous cell vulvar cancer except stage Ia disease regardless of the received treatment
2. Patients with recurrent squamous cell vulvar cancer, if the relapse was not only treated with a surgical excision.
3. Or alternatively, dependent on the decision of the participating center:

   -Patients with primary or relapsed squamous cell vulvar cancer receiving radio- and/or chemotherapy for treatment regardless of nodal involvement.
4. Patients who were diagnosed with and treated for primary or relapsed vulvar cancer between 1998 and 2008
5. Women aged ≥ 18 years

Exclusion Criteria:

1. Patients with benign or precursor lesions (VIN - vulvar intraepithelial neoplasia) of the vulva
2. Patients with non-squamous neoplasia of the vulva (e.g. melanoma)
3. Patients with verrucous vulvar cancer
4. Patients with relapsed squamous cell vulvar cancer only receiving surgical excision for treatment.
5. Patients with secondary cancers if those interfered with the treatment of vulvar disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective, multicenter study is designed to collect tumor characteristics as well as treatment data from patients diagnosed with primary or recurrent squamous cell cancer of the vulva with emphasis on indication and application of radio- and chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 1618 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Determination of several specific characteristics | Data from vulvar cancer pts between 1998 and 2008 will be included in the study. This also includes node negative patients receiving radi
  * Determination of the fraction of node positive patients to estimate the number of participating centers and sample size for a subsequent prospective trial.
  * Determination of the prognostic impact of the number of positive lymph nodes and the stage of disease to define indication criteria for adjuvant radio/chemotherapy for a subsequent prospective trial.
  * Identification of indication criteria for adjuvant/therapeutic/palliative radio/chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Sven Mahner, MD PhD, Principal Investigator — University Medical Center Hamburg-Eppendorf, Department of Gynecology
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Result] Mahner S, Jueckstock J, Hilpert F, Neuser P, Harter P, de Gregorio N, Hasenburg A, Sehouli J, Habermann A, Hillemanns P, Fuerst S, Strauss HG, Baumann K, Thiel F, Mustea A, Meier W, du Bois A, Griebel LF, Woelber L; AGO-CaRE 1 investigators. Adjuvant therapy in lymph node-positive vulvar cancer: the AGO-CaRE-1 study. J Natl Cancer Inst. 2015 Jan 24;107(3):dju426. doi: 10.1093/jnci/dju426. Print 2015 Mar. PMID 25618900